CLINICAL TRIAL: NCT03200145
Title: Residències Centrades en Les Persones (RECENPE): avaluació de l'Impacte d'un Model d'ACP en residències Per Persones Grans
Brief Title: Person Centered Nursing Homes: Impact Assessment Of Centered Person Care In Nursing Homes
Acronym: RECENPE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundacio Salut i Envelliment UAB (Other)
Collaborators: SUMAR empresa d'acció social de Catalunya (Unknown)
Responsible Party: Sponsor
Other Study IDs: FSIE1704; CEEAH - 3786 (Other: Comissió d'Ètica Animal en Experimentació i Humana)
Record Dates: First submitted 2017-06-20; First posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Health Services for the Aged; Quality of Life; Mood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Control: The control group is made by persons living in nursing homes under usual care
  Interventions: Other: ACP intervention

INTERVENTIONS:
Other: ACP intervention — The intervention group made by persons living in nursing homes using a person centered attention model relying on two dimensions:
  1. - Attention to the person based on:
     * Knowledge of the person in several dimensions (biological, psychological, social, etc), interests and preferences.
     * Respect and acknowledge of the person.
     * Promotion of the autonomy.
     * Personalized treatment, with tailored attention and integrative cures
     * Protection of physical well-being, preventing damages and risks and promoting healthy habits.
     * Promotion of independence on daily activities.
     * Protection of privacy and personal matters
  2. - Positive environment based on:
     * Physical space, including accessibility, comfort, homely environment, with stimulating spaces for physical activity, social relationships and significant activities for the persons.
     * Social relationships, with proximity and collaboration with families.
     * Friendly organization, with empathetic professionals empowering users.

SUMMARY:
Cohort Observational Study. The study will assess differences in quality of life, well-being and mood between persons living in a nursing home following usual care and persons living in nursing homes following a centered person care model.

Initially, the follow up will last 6 months, with the possibility to be extended.

ELIGIBILITY:
Inclusion Criteria:

* Persons living in nursing homes
* Consent from the person (or legal representative, if the person is not able)

Exclusion Criteria:

* Terminal illness
* Living temporary in a nursing home

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Persons of any age with or without cognitive impairment living indefinitely in a nursing home
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2017-06-27 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Thriving in nursing homes | 0, 6 months
  Thriving in nursing homes will be assessed with the Thriving of Older People Assessment Scale (TOPAS).
  Investigators will assess the change between groups.
Quality of life | 0, 6 months
  Quality of life will be assessed with the Euroqol 5D-5L. Investigators will assess the change between groups.
Well-being | 0, 6 months
  Well-being will be assessed by the WHO (Five) Well Being Index (1998 version). Investigators will assess the change between groups.

SECONDARY OUTCOMES:
Depressive symptoms | 0, 6 months
  Cognitive impairment affects the assessment of depressive symptoms. For this reason, according to their stage using the Reisberg Global Deterioration Scale, investigators will assess the presence or absence of depressive symptoms with two tools
  * stage 0 to 4: investigators will consider that a person has depressive symptoms with a score of 6 or more using the 15 items Yesavage Geriatric Depression Scale,
  * stage 5 to 7: investigators will consider that a person has depressive symptoms with a score of 11 or more using the Cornell Depression Scale.
  Investigators will assess the change in the prevalence of depressive symptoms between groups.
Neuropsychiatric inventory | 0,6 months
  Neuropsychiatric symptoms will be assessed with the Brief Neuropsychiatric inventory(NPI-Q). Investigators will assess the change between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Rojano Luque, MD, Principal Investigator — Fundació Salut i Envelliment UAB
Locations (2):
- Spain (2):
  - Residència "Casa del Avis", Sant Sadurní d'Anoia, Barcelona
  - Residència i Centre de dia Sant Hilari, Sant Hilari Sacalm, Girona

IPD SHARING:
Plan to Share IPD: Undecided